CLINICAL TRIAL: NCT06223685
Title: Randomized, Double-blind, Placebo-Controlled Study on Efficacy of a Dietary Intervention With Probiotic Bacterial Strains as an Adjunct to Treatment of Small Intestinal Bacterial Overgrowth With Rifaximin
Brief Title: The Efficacy of Probiotics as an Adjunct to Treatment of SIBO With Rifaximin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB-006/15/2023
Record Dates: First submitted 2023-05-24; First posted 2024-01-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-04

CONDITIONS: Irritable Bowel Syndrome; Small Intestinal Bacterial Overgrowth; SIBO
Keywords: SIBO; rifaximin; probiotics; intestinal permeability
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin; Probiotics

STUDY DESIGN:
Intervention Model Description: A prospective randomized, placebo-controlled, double-blinded study of 100 patients with hydrogen-methane breath test-confirmed small intestinal bacterial overgrowth (SIBO) and symptoms, to evaluate the efficacy of a dietary intervention using probiotic bacterial strains as adjunctive therapy to rifaximin.
  Half of patients included in the study according to the standard of therapeutic management of SIBO will receive a prescription for rifaximin at a dose of 1200 mg/d for 14 days (Xifaxan 200 mg, 3 op. of 28 tablets, DS. 3 x 400mg) and the other half will receive a prescription for rifaximin at a dose of 1600 mg/d for 14 days (Xifaxan 200 mg, 4 op. of 28 tablets, DS. 4 x 400mg)
  50 patients will be randomly assigned to an arm receiving a 4enteric probotic, while 50 patients will receive capsules that will have an identical shell to the probiotic, but will contain only potato starch.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Probiotic+Rifaximin 1200mg/day (Experimental): Dosage 2x1 capsule/day. 12 weeks
  Probiotic, which will contain a combination of four freeze-dried strains of probiotic bacteria in DRcaps enteral capsulesTM . These are capsules that protect the probiotics from the effects of hydrochloric acid in the stomach, as they only dissolve in the intestines. The tested composition of probiotics is on sale in Poland, Italy, Taiwan, among other countries. It has a positive recommendation of the Institute "Pomnik-Center for Children's Health" No. 16/DJW/2022.
  (Lactococcus lactis Rosell® - 1058, Lactobacillus casei Rosell® - 215, Lactobacillus helvetius Rosell® - 52, Bifidobacterium bifidum Rosell® - 71) AND Rifaximin at a dose of 1200 mg/d for 14 days (Xifaxan 200 mg, 3 op. of 28 tablets, DS. 3 x 400mg)
  Interventions: Drug: Rifaximin (Xifaxan) 1200mg/day; Dietary Supplement: Probiotic
- Placebo+Rifaximin 1600mg/day (Placebo Comparator): Capsules that look identical to the probiotic and contain potato starch and a shell: hydroxypropylmethylcellulose, gellan gum.
  Dosage 2x1 capsule per day. 12 weeks AND Rifaximin at a dose of 1600 mg/d for 14 days (Xifaxan 200 mg, 4 op. of 28 tablets, DS. 4 x 400mg)
  Interventions: Drug: XIFAXAN® (Rifaximin) 1600mg/day
- Control group (No Intervention): The control group will consist of healthy subjects (25 subjects) without SIBO (with a negative hydrogen-methane test) and without NAFLD (CAP<248dB/m, TE<6.5kPa).
- Probiotic + Rifaximin 1600mg/day (Experimental): Dosage 2x1 capsule/day. 12 weeks
  Probiotic, which will contain a combination of four freeze-dried strains of probiotic bacteria in DRcaps enteral capsulesTM . These are capsules that protect the probiotics from the effects of hydrochloric acid in the stomach, as they only dissolve in the intestines. The tested composition of probiotics is on sale in Poland, Italy, Taiwan, among other countries. It has a positive recommendation of the Institute "Pomnik-Center for Children's Health" No. 16/DJW/2022.
  (Lactococcus lactis Rosell® - 1058, Lactobacillus casei Rosell® - 215, Lactobacillus helvetius Rosell® - 52, Bifidobacterium bifidum Rosell® - 71) AND Rifaximin at a dose of 1600 mg/d for 14 days (Xifaxan 200 mg, 4 op. of 28 tablets, DS. 4 x 400mg)
  Interventions: Dietary Supplement: Probiotic; Drug: XIFAXAN® (Rifaximin) 1600mg/day
- Placebo+Rifaximin 1200mg/day (Placebo Comparator): Capsules that look identical to the probiotic and contain potato starch and a shell: hydroxypropylmethylcellulose, gellan gum.
  Dosage 2x1 capsule per day. 12 weeks AND Rifaximin at a dose of 1200 mg/d for 14 days (Xifaxan 200 mg, 3 op. of 28 tablets, DS. 3 x 400mg)
  Interventions: Drug: Rifaximin (Xifaxan) 1200mg/day

INTERVENTIONS:
Drug: Rifaximin (Xifaxan) 1200mg/day — Dosage 3x2 tablets per day 14 days
  Other Names: Xifaxan
  Arms: Placebo+Rifaximin 1200mg/day; Probiotic+Rifaximin 1200mg/day
Dietary Supplement: Probiotic — 2x1 capsules per day. 12 weeks.
  Arms: Probiotic + Rifaximin 1600mg/day; Probiotic+Rifaximin 1200mg/day
Drug: XIFAXAN® (Rifaximin) 1600mg/day — Dosage 4x2 tablets per day 14 days
  Arms: Placebo+Rifaximin 1600mg/day; Probiotic + Rifaximin 1600mg/day

SUMMARY:
The goal of this clinical trial is to test the effectiveness of probiotic bacterial supplements as an additional therapeutic modality in patients with small intestine bacterial overgrowth who receive oral antibiotic treatment (rifaximin)

The main questions it aims to answer are:

1 To evaluate the effectiveness of a dietary intervention using pro-biotic bacterial strains as an adjunct to treatment of SIBO with rifaximin.

2. Evaluation of ultrasonographic imaging of mesenteric lymph nodes in patients with SIBO.

3. Evaluation of the effect of rifaximin treatment and dietary intervention on non-alcoholic fatty liver disease activity parameters in patients with coexisting NAFLD and SIBO.

According to the study schedule, a total of 3 visits will be made within 3 months. Visit 1, after 6 weeks Visit 2 and after another 6 weeks, Visit 3. Patients will also be invited to a follow-up Visit 4, three months after completing participation in the study.

All study participants will receive treatment recommendations for SIBO in accordance with standard practice - a 14-day antibiotic treatment with Rifaximin.

In addition, a randomly selected half of the study participants will receive probiotic therapy and half a placebo.

* An ultrasound examination of the mesenteric root lymph nodes will be performed at each visit,
* followed by a lier steatosis/fibrosis assessment using SWE elastography or FibroScan.
* Blood sampling is required on each visit. All study participants will receive detailed guidelines during dietary consultations at each visit for the use of a low FODMAP diet.
* Each participant will receive a paper diary on how to assess the severity of bloating and evaluate bowel movements, which must be filled out daily.
* In addition, at the visits the patient will be asked to fill out an additional questionnaire on other gastrointestinal complaints and mental health.

DETAILED DESCRIPTION:
The investigators plan to include 100 participants in the study. The control group will consist of healthy subjects (25 subjects) without SIBO (with a negative hydrogen-methane test) and without NAFLD (CAP<248dB/m, TE<6.5kPa). These patients will have only one visit, at which an abdominal ultrasound will be performed with assessment of mesenteric root lymph nodes, and blood will be drawn for biochemical tests, as well as blood and stool for determination of intestinal barrier integrity markers.

The experiment will be conducted at SONOMED Medical Center from April 2023. until April 2025.

According to the survey scheme, a total of 4 visits will be made during the project. The planned procedures at each visit are outlined below.

Table 1 Scheme of the study Visit 1 (Week 0)

* Ultrasound of the mesenteric root
* SWE elastography, UGAP and Fibroscan (in everyone to identify the subgroup with NAFLD)
* Prescription issue: Xifaxan 1200mg/d for 14 days (3 packs, 28 tablets each)
* Randomization
* drug issue: 4Enteric/Placebo
* Consultation of a nutritionist (issuance of recommendations for stage 1 of the low FODMAP diet)
* anthropometric measurements
* blood draw
* collection of a stool sample
* completion of ailment questionnaires
* Completion of nutrition and physical activity questionnaires
* issuance of SIBO symptom diaries

Visit 2 (Week 6)

* Ultrasound of the mesenteric root,
* SWE elastography + UGAP and Fibroscan (in the subgroup with NAFLD)
* Dietitian consultation (control of low FODMAP diet)
* Implementation of the 2nd stage of the diet
* anthropometric measurements
* blood draw
* collection of a stool sample
* completion of ailment questionnaires
* issuance of SIBO symptom diaries

Visit 3 (Week 12)

* Ultrasound of the mesenteric root
* SWE elastography + UGAP and Fibroscan (in the subgroup with NAFLD)
* Dietitian consultation (control of low FODMAP diet). Implementation of stage 3
* anthropometric measurements
* blood draw
* collection of a stool sample
* completion of ailment questionnaires
* hydrogen-methane test

Follow-up (Week 24)

* SWE elastography + UGAP and Fibroscan (in the subgroup with NAFLD)
* anthropometric measurements
* completion of ailment questionnaires

Method

1. Anthropometric measurements Measurement of height, weight, abdominal circumference, body composition analysis using the Tanita BC-545N impedance scale will be performed on all patients, fasting.
2. Collection of venous blood

   a. Biochemical tests (15 ml of venous blood; fasted) All included patients will undergo a standard panel of biochemical tests to assess liver function and metabolism (including AST, ALT, GGTP, triglycerides, total cholesterol and its HDL fractions. LDL, glucose, HOMA-IR, CRP). In all patients, serum will also be secured and stored for the determination of pro-inflammatory cytokines (TNF-α, IL-1β, IL-6, IL-8, IFN-γ) and in patients with pathological lymph nodes for the determination of fibrogenesis indicators (TGF-β, TIMP-1, PIIINP, PINP, collagen IV) and IgG4 antibodies.

   Metabolomic analysis (untargeted metabolome, short-chain fatty acids, trimethylamines, trimethylamine oxide, indoxyl sulfate, tryptophan catabolites) will be performed on a quadrupole mass spectrometer coupled to a time-of-flight (QTOF) analyzer coupled to a high-performance liquid chromatograph (UHPLC) from AB Sciex - TripleTOF® 6600+.

   Data analysis will be carried out by metabolomic analysis system - XCMSplus.

   c. Study of markers of intestinal barrier damage in blood (4 ml of venous blood per clot) Plasma indicators of intestinal barrier damage will be determined in all included patients: intestinal fatty-acid binding protein (I-FABP ), calprotectin

   Description of the procedure for preparing the material:

   i. After the blood is drawn, it is being set aside for about 30-60 minutes ii. Spinning - 5 minutes at 3500-4000 rpm, iii. Extract serum and collect into 3-4 tubes (standard 1.5-2ml) of 500ul (1 tube for each protein)
3. collection of 2 stool samples Each patient will be asked to collect biological material using the Forged kit (https://www.fecesvanger.nl/en_GB/c-2866881/product-info/). Metabolomic tests and determination of markers of intestinal barrier damage will be performed from the collected stool samples.

   The procedures for developing the 16S sequences follow the protocols used during the Earth Microbiome Project. Bioinformatics analysis will be performed using the QIIME tool. Operational taxonomic units (OTUs, sOTUs) are determined using two alternative methods (pipelines, algorithms).
   1. Fecal metabolomics test Metabolomic analysis (untargeted metabolome, short-chain fatty acids, trimethylamines, trimethylamine oxide, indoxyl sulfate, tryptophan catabolites) will be performed on a quadrupole mass spectrometer coupled to a time-of-flight (QTOF) analyzer coupled to a high-performance liquid chromatograph (UHPLC) from AB Sciex - TripleTOF® 6600+.

      Data analysis will be carried out by metabolomic analysis system - XCMSplus.
   2. Study of markers of intestinal barrier damage in feces: IFAB-P, zonulin, calprotectin
4. Questionnaires:

   1. regarding SIBO related ailments I. Diary of symptoms in a patient with SIBO (Appendix 1) Assessment of bloating severity based on the VAS scale and assessment of bowel movements based on the Bristol stool scale. The Visual Analog Scale (VAS) is a tool used for subjective assessment of pain. The VAS scale consists of a line 100 mm long, with two endpoints indicating 0 ("no bloating") and 100 ("unbearable bloating"). The patient is asked to mark on the line the intensity of the bloating he or she is experiencing.

      The Bristol Stool Form Scale (BSFS) is used to assess bowel passage and stool shape and consistency. It includes 7 basic types of stool that help estimate the regularity of bowel movements.

      II. GSRS scale (Appendix 2) The Gastrointestinal Symptom Rating Scale (GSRS) questionnaire assesses the severity and frequency of symptoms over the past week and their impact on daily functioning. It consists of 15 questions, relating to 5 general symptoms found in gastrointestinal diseases. Questions are scored using a 7-point Likert scale, where 1 indicates the absence of troublesome symptoms and 7 indicates the presence of very troublesome symptoms. The higher the total score obtained, the greater the severity of the symptoms.

      III. PHQ-9 The PHQ-9 Patient Health Questionnaire (PHQ-9) is designed to screen for depression, and is used in the initial diagnosis.
   2. Regarding Nutrition and Physical Activity I. FFQ Questionnaire collecting dietary data from the last 12 months preceding the survey II. The Godin Leisure Time Exercise Questionnaire (The Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ) The GLTEQ (shortened to GSLTPAQ) is one of the most widely used scales to measure physical activity.
5. mesenteric root ultrasound The examination will be carried out in all project participants by a specialist in internal medicine certified by the PTU to perform ultrasound, with the help of an Aixplorer ultrasound machine (SuperSonic Imagine) using a linear L18-5 or convex C6-1X type head.
6. non-invasive assessment of liver fibrosis and steatosis (in all, to identify a subgroup with NAFLD)

   1. SWE elastography The research will be performed with an Aixplorer from SuperSonic Imagine using a Convex C6-1X type head in SWE (shear wave elastography) mode by the Principal Investigator.
   2. UGAP In the ultrasound-guided attenuation parameter (UGAP) system, attenuation is quantified and represented by a color map in a real-time B-type presentation.
   3. Fibroscan Non-invasive measurement of the degree of liver fibrosis will be performed with the FibroScan device by the Principal Investigator.
   4. Hydrogen-methane breath test The tests will be performed using Quintron's BreathTracker S.C. hydrogen and methane analyzer.

According to the guidelines of the American College of Gastroenterology (ACG), a positive hydrogen test result is considered a rise of ≥ 20 ppm from baseline to the 90th minute of the test. A positive methane test result is considered an increase of ≥ 10 ppm at any time during the breath test.

7. treatment/intervention

1. rifaximin 1200 mg/d for 14 days (3 op. a 28 tablets) - all patients

   All patients included in the study according to the standard of therapeutic management of SIBO will receive a prescription for rifaximin at a dose of 1200 mg/d for 14 days (Xifaxan 200 mg, 3 op. of 28 tablets, DS. 3 x 400mg). According to the SmPC, rifaximin is registered in Poland for the treatment of gastrointestinal diseases such as intestinal infections, which is bacterial overgrowth of the small intestine. The suggested dose ranges from 200 mg (1 tablet) every 8 hours to 400 mg (2 tablets) every 8-12 hours. According to the American College of Gastroenterology (ACG) guidelines, it is the suggested antibiotic for the treatment of SIBO, and the efficacy of therapy with rifaximin at a dose of 550 mg three times a day is estimated at 61-78%. It is a semi-synthetic derivative of rifamycin SV, occurs in the α polymorphic form, has a bactericidal effect, and is practically not absorbed from the gastrointestinal tract. The mechanism of action is based on irreversible binding of rifaximin to the β subunit of DNA-dependent RNA polymerase and, as a result, inhibition of bacterial RNA and protein synthesis. Rifaximin exhibits a broad spectrum of antimicrobial activity, including most Gram-positive and Gram-negative, aerobic and anaerobic bacteria, including ammonia-producing species. It can inhibit the proliferation of bacteria that cause urea deamination, thereby reducing the production of ammonia and other substances thought to play an important role in the pathogenesis of hepatic encephalopathy. It acts topically rather than systemically. It is counted among the eubiotics, which are types of antimicrobial drugs that, when introduced into the body, change the composition of the intestinal microflora. The number of side effects is small, hence rifaximin is considered a safe, well-studied and highly effective drug.

   Contraindications: Hypersensitivity to rifaximin or other rifamycins, or to any of the excipients. Hypersensitivity reactions include exfoliative dermatitis, angioedema and anaphylaxis. Intestinal obstruction, even partial, and severe ulcerative intestinal damage.
2. randomization: probiotic/placebo release Probiotic, which will contain a combination of four freeze-dried strains of probiotic bacteria in DRcaps enteral capsulesTM . These are capsules that protect the probiotics from the effects of hydrochloric acid in the stomach, as they only dissolve in the intestines. The tested composition of probiotics is on sale in Poland, Italy, Taiwan, among other countries. It has a positive opinion of the Institute "Pomnik-Center for Children's Health" No. 16/DJW/2022. The composition in the table below. Dosage 2x1 capsule per day.

   Placebo Capsules that look identical to the probiotic and contain potato starch and a shell: hydroxypropylmethylcellulose, gellan gum.
3. Dietitian consultation and issuance of recommendations on low FODMAPs diet The low-FODMAPs diet (LFD) is an elimination protocol based on temporarily limiting the intake of highly fermentable substances such as fructooligosaccharides, oligosaccharides, disaccharides, monosaccharides and polyols.

Conditions for discontinuing a medical experiment The subject conducting the experiment is obliged to discontinue it if, during the course of the experiment, there is a risk to the participant's health that exceeds the expected benefits. The person participating in the experiment may at any time (at any stage of the experiment) revoke the previously given consent without giving a reason. Then the entity conducting the experiment is obliged to stop it.

ELIGIBILITY:
Inclusion Criteria:

* positive hydrogen OR methane breath test
* SIBO symptoms seen as:

moderate or severe bloating for at least 50% of days in the past 3 months if hydrogen test (+) OR constipation (< 3 bowel movements/week) in the past 3 months if methane test (+)

Exclusion Criteria:

* age <18
* age >70,
* current proton pump inhibitor therapy,
* antibiotic therapy in the past 3 months,
* probiotic therapy in the past 2 weeks,
* daily intake of >30 g of ethanol for men
* daily intake of >20 g of ethanol for women,
* hepatitis B or C virus infection,
* other liver disease,
* celiac disease,
* severe chronic disease (m.e.g. chronic kidney disease, congestive heart failure, cancer, liver failure),
* current symptoms of acute infection,
* pregnancy,
* vegan diet or following non-recommended diets such as ketogenic,
* patients with very high physical activity (> 5 x week of 100 min of strength training).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change in bloating on Visual Analog Score | 12 weeks
  Visual Analog Score (range 0-10, the lower the better) reduction in bloating by 50% in patients with a baseline positive hydrogen test
Change in bowel movements in a bowel-movement diary | 12 weeks
  increase in bowel frequency by 1/week in patients with a baseline positive methane test

SECONDARY OUTCOMES:
The number of patients with a negative hydrogen test | 12 weeks
  < 20 ppm in 90 minutes in hydrogen test
The number of patients with a negative methane test | 12 weeks
  no increase ≥ 10 ppm in 90 minutes in methane test)
Change in subjective symptoms on Visual Analog Score | 12 weeks
  assessed by VAS - bloating and abdominal pain or discomfort (range 0-10, the lower the better)
Change in subjective symptoms on Gastrointestinal Symptom Rating | 12 weeks
  change in symptoms expressed as a decrease in total score on the GSRS (range 1-7, the lower score the better)
Change in patient-reported stool quality by Bristol Stool Chart | 12 weeks
  Range 1-7 Types 1 and 2 indicate severe or mild constipation, 3 and 4 - normal stool 5 indicating lack of dietary fiber, 6 and 7 indicate mild or severe diarrhoea.
Depression risk in Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
  Range 0-27 points Interpretation: Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Change in mesenteric root lymph node ultrasound | 12 weeks
  reduction of peri-nodal inflammation and reduction/atrophy of mesenteric root lymph nodes is a favorable outcome
Improved indices of liver function and metabolism | 12 weeks
  as well as inflammatory markers (blood biochemical tests)
Changes in liver tests - alanine transaminase (ALT) | 12 weeks
  normal range 7 to 56 U/L (units per liter)
Changes in liver tests - aspartate transaminase (AST) | 12 weeks
  normal range 8 to 33 U/L (units per liter)
Changes in liver tests - Gamma-glutamyl transpeptidase (GGTP or GGT) | 12 weeks
  7 to 47 U/L for males. 5 to 25 U/L for females. (units per liter)
Changes in liver tests - triglycerides | 12 weeks
  Normal - Less than 150 milligrams per deciliter (mg/dL), or less than 1.7 millimoles per liter (mmol/L) Borderline high - 150 to 199 mg/dL (1.8 to 2.2 mmol/L) High - 200 to 499 mg/dL (2.3 to 5.6 mmol/L)
Changes in cholesterol | 12 weeks
  A total cholesterol level of less than 200 mg/dL (5.17 mmol/L) is normal.
Changes in liver function - Fatty Liver Index | 12 weeks
  Fatty Liver Index (FLI) is calculated using a formula which requires patient's triglycerides, BMI, GGT and waist circumference
  FLI = (e0.953×loge(triglycerides)+0.139×BMI+0.718×loge(GGT)+0.053×waistcircumference-15.745)/ (1 + e0.953×loge(triglycerides)+0.139×BMI+0.718×loge(GGT)+0.053×waistcircumference-15.745) × 100.
  FLI <30 most likely excludes fatty liver disease. FLI ≥60 confirms the presence of disease
Changes in the microbiome and metabolome | 12 weeks
  qualitative microbiota assessment based on stool and blood samples
Change in intestinal permeability parameters - intestinal fatty acid binding protein | 12 weeks
  Normal range values have not been well validated. Generally lower value at the end of treatment is considered a favorable outcome
Change in intestinal permeability parameters - calprotectin | 12 weeks
  Normal range values have not been well validated. Generally lower value at the end of treatment is considered a favorable outcome
Change in intestinal permeability parameters - fecal zonulin content | 12 weeks
  Normal range values have not been well validated.
Change of hepatic steatosis - Controlled Attenuation Parameter | 12 weeks
  assessed with Fibroscan. Lower values of CAP at the end of treatment indicate steatosis reduction.
Change of hepatic steatosis - Ultrasound-Guided Attenuation Parameter | 12 weeks
  assessed with ultrasound. Lower values of UGAP at the end of treatment indicate steatosis reduction.
Change of hepatic fibrosis - Shear Wave Elastography | 12 weeks
  assessed with ultrasound. Lower values of SWE at the end of treatment indicate fibrosis reduction.
Change of hepatic fibrosis - Transient Elastography | 12 weeks
  assessed with Fibroscan. Lower values of TE at the end of treatment indicate fibrosis reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Kozlowska-Petriczko, MD, PhD, Principal Investigator — Pomeranian Medical University
Locations (1):
- Sonomed CENTRUM MEDYCZNE, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No